CLINICAL TRIAL: NCT06715722
Title: Comparison of Abutments Engagement Configurations in Implant Supported Fixed Partial Dentures: a Randomized Clinical Trial
Brief Title: Comparison of Abutments Engagement Configurations in Implant Supported Fixed Partial Dentures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Mohammad AL-Rababáh, Associate Professor, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10/2024/28042
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Dental Implant
Keywords: Implant abutment connection; Dental implant; Fixed dental prosthesis; Engaging abutment; Non-engaging abutment; Conical connections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking Description
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- hexed non hexed (Experimental): a 3-unit screw-retained implant bridge over two conical internal hex implants will be supported using hexed and non hexed abutments
  Interventions: Device: hexed non hexed
- non hexed non hexed (Active Comparator): a 3-unit screw-retained implant bridge over two conical internal hex implants will be supported using two non-hexed abutments
  Interventions: Device: non-hexed non-hexed

INTERVENTIONS:
Device: hexed non hexed — A 3-unit screw-retained implant bridge over two conical internal hex implants will be supported using one hexed and one non-hexed abutment.
  Arms: hexed non hexed
Device: non-hexed non-hexed — a 3-unit screw-retained implant bridge over two conical internal hex implants will be supported using two non-hexed abutments
  Arms: non hexed non hexed

SUMMARY:
This study focuses on the comparison of different implant abutment connections configurations in implant supported screw retained fixed dental prostheses assessing their clinical and radiographic outcomes and to evaluate which implant abutment connection configuration have less biological and technical complications.

DETAILED DESCRIPTION:
Study design:

This study is designed as a parallel group randomized controlled trial with an allocation ratio of 1:1.

The (PICO) study design: population will be patients from Jordan University Hospital aged 18 years or older, patients who will receive 2 internal connection dental implants to replace 3 posterior missing teeth in the mandible with a 3 unit screw-retained FDP with sufficient bone volume and controlled oral hygiene. The intervention group will receive a screw-retained FDP with conical engaging and non engaging abutment configuration, while the comparator group will a screw-retained FDP with both conical non engaging abutment configuration. The primary outcome is changes in marginal bone levels, and the secondary outcomes include technical and mechanical complications, biological complications, and patient satisfaction.

Both groups will receive 2 internal connection implants in the posterior mandible in healed sites of at least 3 months (guided implant surgery). The surgical procedure will follow standardized protocols, with no variations between groups other than the types of implant abutment connections used.

Blinded assessors will perform radiographic and clinical evaluations at designated follow-up visits: definitive loading, after 6 months of loading, after 2 years loading.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with edentulous span in the posterior mandible of 3 missing teeth.
* Candidates for an implant supported FDP in the posterior mandible.
* Teeth in area of interest extracted at least 3 months prior.
* Bone grafting not needed or only minor GBR needed.
* Controlled oral hygiene.
* Sufficient bone volume.

Exclusion Criteria:

* Patients with edentulous span of less than 3 missing teeth (not eligible to receive a 3 unit 2 implant supported FDP)
* Patients with healing period of extraction sites less than 3 months.
* Extensive bone grafting required prior to or during implant placement.
* Active Bruxism.
* Heavy smoker (> 10 cigarettes).
* Systemic diseases that might affect bone healing.
* Patients who are not willing or unable to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-11-10 (Estimated)

PRIMARY OUTCOMES:
Marginal Bone Loss | Baseline (day of definitive loading) and at 1-year follow-up post-loading.
  Marginal bone level changes by standardized periapical radiographs.

SECONDARY OUTCOMES:
Technical or mechanical complications | 1 year
  screw loosening, screw fracture, abutment or implant fracture, prosthesis fracture or chipping
Biological complications | 1 year
  Peri implant bone loss, early implant failure.
Patient satisfaction | 1 year
  To be assesses by oral health impact profile-14 (OHIP-14), The scale includes 14 items covering various aspects of oral health-related quality of life, Score Range: from 0 to 56, Higher OHIP-14 scores indicate a worse outcome, representing a greater negative impact of oral health issues on quality of life, while lower scores suggest a better outcome or less impact on the individual's daily life.

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No